CLINICAL TRIAL: NCT00782860
Title: Early Pregnancy Failure: Factors Affecting Successful Medical Termination Treatment
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Other Study IDs: 03-08-2008
Record Dates: First submitted 2008-10-28; First posted 2008-10-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Early Pregnancy Failure
Keywords: Early pregnancy failure; Misoprostol; Gestational sac volume

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- unsuccessful termination: unsuccessful termination of early pregnancy failure with Misoprostol
- successful termination: successful termination of early pregnancy failure with Misoprostol

SUMMARY:
The main purpose of our study was to which determine factors, those measured by ultrasound and also demographic and clinical factors (age, number of previous pregnancies, abortions and deliveries) predict outcome of medical treatment for early pregnancy failure. Our hypothesis was that gestational sac volume predicts outcome of medical treatment for early pregnancy failure.

ELIGIBILITY:
Inclusion Criteria:

* Crown rump length (CRL) is appropriate to less than 12 weeks.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with missed abortion or anembryonic pregnancy, with existing intrauterine pregnancy sac
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
An empty uterus or an endometrial lining with thickness of less than 30mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital-Nahariya, Nahariya, Israel